CLINICAL TRIAL: NCT00974363
Title: Persistence of Antibodies After Vaccination With GSK Biologicals' Meningococcal Vaccine GSK134612 in Adolescents and Young Adults
Brief Title: Study to Evaluate Persistence of Antibodies After Vaccination With Meningococcal Vaccine GSK 134612
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112148
Record Dates: First submitted 2009-09-07; First posted 2009-09-10 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2016-12

CONDITIONS: Infections, Meningococcal
Keywords: meningococcal vaccine GSK 134612
MeSH Terms: conditions — Meningococcal Infections | interventions — Blood Specimen Collection

ARMS (2):
- Group A (Experimental): Subjects who received GSK Biologicals' meningococcal vaccine 134612 in the primary vaccination study 109069.
  Interventions: Procedure: Blood Sampling
- Group B (Active Comparator): Subjects who received MencevaxTM ACWY in the primary vaccination study 109069.
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — A blood sample will be taken yearly at each long-term follow-up visit (i.e. Year 2 through Year 5) after vaccination during the primary study. No vaccines are administered in the long-term follow-up study

SUMMARY:
Subjects were previously vaccinated at 11 to 17 years of age. This extension phase starts 24 months after vaccination and the subjects who were vaccinated in the primary study will be enrolled in this extension phase. No new subjects will be enrolled.

DETAILED DESCRIPTION:
Subjects were previously vaccinated at 11 to 17 months of age with GSK Biologicals' meningococcal vaccine 134612 or with Mencevax™. This extension phase starts 24 months after vaccination and the subjects who were vaccinated in the primary study will be enrolled in this extension phase. No new studies will be enrolled. The subjects will have 4 blood samples taken: at 24, 36, 48 and 60 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s)/guardian(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female having been vaccinated with a meningococcal vaccine in the primary study 109069.
* Written informed consent obtained from parent(s)/guardian(s) of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject has achieved the 18th birthday.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the subject's first visit.
* History of meningococcal disease; such cases will be documented.
* Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine since previous vaccination in study 109069.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Administration of immunoglobulins and/or any blood products within the three months preceding the subject's first visit.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy
* Subjects who withdrew consent to be contacted for follow-up studies.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 697 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- India (4):
  - GSK Investigational Site, Goa
  - GSK Investigational Site, Indore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- GSK Investigational Site, City of Muntinlupa, Philippines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 697 subjects enrolled in this study, only 689 were vaccinated and hence started the study.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix™ Group: Healthy adolescents and young adults between and including 11 to 17 years of age, who were previously vaccinated in the primary study MenACWY-TT-036 (109069) with a single dose of Nimenrix™ (MenACWY-TT) vaccine, intramuscularly into the deltoid region of the non-dominant arm.
- Mencevax™ Group: Healthy adolescents and young adults between and including 11 to 17 years of age, who were previously vaccinated in the primary study MenACWY-TT-036 (109069) with a single dose of Mencevax™ (MenACWY) vaccine, intramuscularly into the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Started | 521 | 168
Completed | 521 | 168
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix™ Group | Mencevax™ Group | Total
Number analyzed (Participants) | 521 | 168 | 689
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.4 (1.94) | 16.4 (2) | 16.4 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 86 | 359
  Male | 248 | 82 | 330

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against the Vaccine Meningococcal Serogroups
Description: A seroprotected subject was defined as a subject who had anti-meningococcal serogroups A (MenA), C (MenC), W-135 (MenW-135) and Y (MenY) antibody titers equal to or above (≥) the cut-off value of 1:8. The persistence of serum bactericidal antibodies was evaluated using baby rabbit complement (rSBA) titers. The blood analyses were performed at the GSK Biologicals' laboratory.
Time Frame: At Month 24 post primary dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for persistence, which included all evaluable subjects for whom assay results were available for at least one tested antigen.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 407 | 132
Subjects
  rSBA- MenA, GSK laboratory [N=405;132] | 404 | 132
  rSBA- MenC, GSK laboratory [N=407;132] | 404 | 131
  rSBA- MenW-135, GSK laboratory [N=407;131] | 405 | 124
  rSBA- MenY, GSK laboratory [N=407;130] | 407 | 126

2. Primary Outcome: Number of Seroprotected Subjects Against the Vaccine Meningococcal Serogroups
Description: A seroprotected subject was defined as a subject who had anti-meningococcal serogroups A (MenA), C (MenC), W-135 (MenW-135) and Y (MenY) antibody titers equal to or above (≥) the cut-off value of 1:8. The persistence of serum bactericidal antibodies was evaluated using baby rabbit complement (rSBA) titers. The blood analyses for this timepoint were performed solely at the Public Health of England's (PHE) laboratory.
Time Frame: At Month 36 post primary dose
Population: The analysis was performed on the ATP cohort for persistence, which included all evaluable subjects for whom assay results were available for at least one tested antigen.
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 449 | 150
Subjects
  rSBA-MenA, PHE laboratory | 417 | 124
  rSBA-MenC, PHE laboratory | 409 | 129
  rSBA-MenW-135, PHE laboratory | 368 | 45
  rSBA-MenY, PHE laboratory | 418 | 87

3. Primary Outcome: Number of Seroprotected Subjects Against the Vaccine Meningococcal Serogroups
Description: as for outcome 2
Time Frame: At Month 48 post primary dose
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 391 | 130
Subjects
  rSBA-MenA, PHE laboratory [N=391;130] | 353 | 105
  rSBA-MenC, PHE laboratory [N=390;130] | 367 | 113
  rSBA-MenW-135, PHE laboratory [N=390;130] | 301 | 35
  rSBA-MenY, PHE laboratory [N=389;130] | 348 | 63

4. Primary Outcome: Number of Seroprotected Subjects Against the Vaccine Meningococcal Serogroups
Description: as for outcome 2
Time Frame: At Month 60 post primary dose
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 236 | 86
Subjects
  rSBA-MenA, PHE laboratory [N=236;86] | 230 | 80
  rSBA-MenC, PHE laboratory [N=236;85] | 209 | 74
  rSBA-MenW-135, PHE laboratory [N=236;86] | 203 | 30
  rSBA-MenY, PHE laboratory [N=236;86] | 228 | 57

5. Secondary Outcome: Number of Seropositive Subjects Against the Vaccine Meningococcal Serogroups
Description: A seropositive subject was defined as a subject who had the anti-meningococcal serogroups A (MenA), C (MenC), W-135 (MenW-135) and Y (MenY) antibody titers equal to or above (≥) the cut-off value of 1:128. The persistence of serum bactericidal antibodies was evaluated using baby rabbit complement (rSBA) titers. The blood analyses were performed at the Public Health of England's (PHE) laboratory and at GSK Biologicals' laboratory.
Time Frame: At Months 24, 36, 48 and 60 post primary dose
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 449 | 150
Subjects
  rSBA-MenA, M24, GSK laboratory [N=405;132] | 403 | 128
  rSBA-MenA, M36, PHE laboratory [N=449;150] | 398 | 118
  rSBA-MenA, M48, PHE laboratory [N=391;130] | 335 | 99
  rSBA-MenA, M60, PHE laboratory [N=236;86] | 219 | 71
  rSBA-MenC, M24, GSK laboratory [N=407;132] | 396 | 125
  rSBA-MenC, M36, PHE laboratory [N=449;150] | 380 | 117
  rSBA-MenC, M48, PHE laboratory [N=390;130] | 347 | 104
  rSBA-MenC, M60, PHE laboratory [N=236;85] | 188 | 68
  rSBA-MenW-135, M24, GSK laboratory [N=407;131] | 403 | 113
  rSBA-MenW-135, M36, PHE laboratory [N=449;150] | 350 | 36
  rSBA-MenW-135, M48, PHE laboratory [N=390;130] | 284 | 25
  rSBA-MenW-135, M60, PHE laboratory [N=236;86] | 195 | 26
  rSBA-MenY, M24, GSK laboratory [N=407;130] | 407 | 123
  rSBA-MenY, M36, PHE laboratory [N=449;150] | 401 | 77
  rSBA-MenY, M48, PHE laboratory [N=389;130] | 333 | 60
  rSBA-MenY, M60, PHE laboratory [N=236;86] | 225 | 56

6. Secondary Outcome: Antibody Titers Against the Vaccine Meningococcal Serogroups
Description: Seropositivity status was defined as the anti-meningococcal serogroups A (MenA), C (MenC), W-135 (MenW-135) and Y (MenY) titers equal to or above the cut-off value of 1:128. Antibody titers were presented as geometric mean titers (GMTs). The blood analyses were performed at the Public Health of England's (PHE) laboratory and at GSK Biologicals' laboratory.
Time Frame: At Months 24, 36, 48 and 60 post primary dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 449 | 150
Titers
  rSBA-MenA, M24, GSK laboratory [N=405;132] | 1493.4 [1369 to 1629] | 780.3 [665.3 to 915.2]
  rSBA-MenA, M36, PHE laboratory [N=449;150] | 448.3 [381.4 to 527.1] | 206 [147.4 to 288.1]
  rSBA-MenA, M48, PHE laboratory [N=391;130] | 386.9 [321.2 to 466.2] | 174.4 [121.2 to 250.8]
  rSBA-MenA, M60, PHE laboratory [N=236;86] | 643.8 [530.7 to 781] | 296 [202.4 to 432.9]
  rSBA-MenC, M24, GSK laboratory [N=407;132] | 1137.5 [1006.1 to 1286] | 1543 [1145.8 to 2077.7]
  rSBA-MenC, M36, PHE laboratory [N=449;150] | 371.4 [309.4 to 445.8] | 389.8 [262 to 579.9]
  rSBA-MenC, M48, PHE laboratory [N=390;130] | 378.5 [319.7 to 448.1] | 364 [242.7 to 545.9]
  rSBA-MenC, M60, PHE laboratory [N=236;85] | 248.6 [194.2 to 318.2] | 366.5 [224.1 to 599.4]
  rSBA-MenW-135, M24, GSK laboratory [N=407;131] | 1977.6 [1775 to 2203.4] | 418.2 [317.6 to 550.6]
  rSBA-MenW-135, M36, PHE laboratory [N=449;150] | 338 [268.4 to 425.6] | 16 [10.9 to 23.6]
  rSBA-MenW-135, M48, PHE laboratory [N=390;130] | 209.8 [163.9 to 268.6] | 11.7 [8.2 to 16.8]
  rSBA-MenW-135, M60, PHE laboratory [N=236;86] | 436.9 [324.4 to 588.4] | 19.7 [11.8 to 32.9]
  rSBA-MenY, M24, GSK laboratory [N=407;130] | 3502.5 [3203.2 to 3829.7] | 1028.3 [797.3 to 1326.1]
  rSBA-MenY, M36, PHE laboratory [N=449;150] | 740.5 [620 to 884.3] | 69.6 [44.6 to 108.6]
  rSBA-MenY, M48, PHE laboratory [N=389;130] | 533.4 [430 to 661.7] | 49.8 [30.7 to 80.9]
  rSBA-MenY, M60, PHE laboratory [N=236;86] | 1000.2 [824.1 to 1214] | 124.9 [71.2 to 219.3]

7. Secondary Outcome: Number of Subjects With Antibody Concentrations Against the Vaccine Polysaccharides
Description: Antibody concentrations against polysaccharide A (anti-PSA), polysaccharide C (anti-PSC), polysaccharide W-135 (anti-PSW-135) and polysaccharide Y (anti-PSY) assessed were equal to or above (≥) the cut-off values of 0.3 micrograms/milliliter (µg/mL ) and 2.0 micrograms/milliliter (µg/mL). Concentration of antibodies was determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: At Month 24 post primary dose
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 208 | 66
Subjects
  Anti-PSA ≥ 0.3 µg/mL, [N=196; 65] | 196 | 65
  Anti-PSA ≥ 2.0 µg/mL, [N=196; 65] | 179 | 64
  Anti-PSC ≥ 0.3 µg/mL, [N=192; 66] | 176 | 66
  Anti-PSC ≥ 2.0 µg/mL, [N=192; 66] | 96 | 62
  Anti-PSW-135 ≥ 0.3 µg/mL, [N=198; 62] | 187 | 61
  Anti-PSW-135 ≥ 2.0 µg/mL, [N=198; 62] | 127 | 49
  Anti-PSY ≥ 0.3 µg/mL, [N=208; 65] | 203 | 63
  Anti-PSY ≥ 2.0 µg/mL, [N=208; 65] | 130 | 51

8. Secondary Outcome: Antibody Concentrations Against the Vaccine Polysaccharides
Description: as for outcome 7
Time Frame: At Month 24 post primary dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Number analyzed (Participants) | 208 | 66
μg/mL
  Anti-PSA [N=196; 65] | 10.16 [8.47 to 12.2] | 18.17 [13.33 to 24.77]
  Anti-PSC [N=192;66] | 1.95 [1.61 to 2.35] | 10.88 [8.22 to 14.41]
  Anti-PSW-135 [N=198;62] | 3.29 [2.71 to 4] | 5.22 [3.74 to 7.27]
  Anti-PSY [N=208;65] | 3.63 [3 to 4.4] | 6.99 [4.83 to 10.11]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): up to Month 24, 36, 48 and 60 post primary vaccination.
Description: No information about unsolicited AEs was collected during this study as no product was administered.
Arm/Group | Nimenrix™ Group | Mencevax™ Group
Serious Adverse Events (participants affected / at risk) | 0/521 | 0/168
Other Adverse Events (participants affected / at risk) | 0/521 | 0/168

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.